CLINICAL TRIAL: NCT02793362
Title: Measurement of Sarcopenia at Post-stroke Rehabilitation Outcome
Status: Completed | Type: Observational
Sponsor: Bucheon St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Geun-Young Park, MD, PhD, Bucheon St. Mary's Hospital
Other Study IDs: HC16OIS0028
Record Dates: First submitted 2016-05-30; First posted 2016-06-08 (Estimated); Last update posted 2019-01-03 (Actual); Status verified 2019-01

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Normal subjects without stroke: 1. subjects who can walk independent without any difficult
  2. subjects without history of CNS or PNS lesion
  3. Modified ranking scale (MRS) <=2
  4. Functional ambulation category (FAC) >=2
- Post stroke patients with sarcopenia(by sarcopenia index): Existence of sarcopenia will be determined by DEXA scan where sarcopenia index of male less than 7.40 kg/m2, that of female less than 5. 14 kg/m2 are considered as sarcopenia.
- Post stroke patients without sarcopenia(by sarcopenia index): patients who do not satisfy the value of DEXA scan where sarcopenia index of male less than 7.40 kg/m2, that of female less than 5. 14 kg/m2 are considered as sarcopenia.
- Post stroke patients with sarcopenia(by lean body mass): Existence of sarcopenia will be determined by DEXA scan where appendicular lean mass less than <19.75 kg in men, and <15.02 kg in women are considered sarcopenia.
- Post stroke patients without sarcopenia(by lean body mass): patienst who do not satisfy the value of DEXA scan where appendicular lean mass less than <19.75 kg in men, and <15.02 kg in women are considered sarcopenia.

SUMMARY:
The purposes of this study are

1. To explore effect of sarcopenia on recovery of post stroke hemiplegia
2. To explore the effect of stroke on sarcopenia and relationship between the degree of sarcopenia and respiration and swallowing function
3. To quantify and qualify post stroke loss of muscle mass
4. To validity the use of echointensity and elastography in evaluation of sarcopenia.

By reaching the above list purposes, sarcopenia can be viewed as one of serious post stroke complications that is closely related to worth functional outcome, thereby emphasizing the importance of evaluation of sarcopenia as well as its prevention.

DETAILED DESCRIPTION:
Sarcopenia occurs frequently among old population. The changes can rather occur earlier after trauma or generalized illness. However, the nature of these sarcopenia is different from that of geriatric population. Post stroke sarcopenia is underestimated however reduction in the motor uni number begins within 4 hours post stroke and after 3 weeks, sarcopenia can be seen in both hemiplegia and normal side. This muscular weakness can hinder functional recovery process.

ELIGIBILITY:
Inclusion Criteria for stroke patients

* First ever subacute stroke patients whose lesions were confirmed in brain imaging (MRI/CT)
* Patients who did not have difficulty in premorbid ambulation or activities of daily living.
* Patients who can follow 1 step obey
* Patients who can perform hand function test
* Patients whose laboratory tests, neurologic, cognitive, and dysphagia evaluations are completed within 1 month from the onset date.
* Patients who admitted/transferred into our department for at least 4 weeks, following conventional rehabilitation protocols.
* Patients with at least 2 of MRS(Modified Ranking Score) and FAC(Functional ambulation category) scores.

Exclusion Criteria: for stroke patients

* Patients who do not meet the above listed criteria
* Patients with double hemiplegia
* Patients with other systemic diseases that can affect loss of muscle mass or causr malnutrition. (Example : chronic inflammatory disease, autoimmune disease, chronic intestinalis, active tuberculosis, immunocompromised state, AIDS, malignancy, pregnancy, amputation, or operation.
* Patients with joint contracture who are difficult to perform sonographic evaluation.
* Traumatic brain injury patients.

Inclusion Criteria for normal subjects

* Subjects who can walk independent without any difficult
* Subjects without history of CNS or PNS lesion
* MRS(Modified ranking scale) <=2
* FAC(functional ambulation category) >=2

Exclusion Criteria for normal subjects

* Patients with other systemic diseases that can affect loss of muscle mass or causr malnutrition. (Example : chronic inflammatory disease, autoimmune disease, chronic intestinalis, active tuberculosis, immunocompromised state, AIDS, malignancy, pregnancy, amputation, or operation.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruited subjects will be allocated into 3 different groups.
  1. Normal subjects without stroke (30 healthy volunteers)
  2. Post stroke patients with sarcopenia (40 first ever stroke patients who admitted to Bucheon St. Mary's Hospital)
  3. Post stroke patients without sarcopenia (40 first ever stroke patients who admitted to Bucheon St. Mary's Hospital)
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2016-05; Primary Completion 2017-05-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Change in K-MBI score from initial evaluation to the final evaluation | 8 weeks, 12 weeks, 16 weeks from the first onset of the stroke

SECONDARY OUTCOMES:
Change in Berg balance scale from initial evaluation to the final evaluation | 8 weeks, 12 weeks, 16 weeks from the first onset of the stroke
Change in Fatigue scale from initial evaluation to the final evaluation | 8 weeks, 12 weeks, 16 weeks from the first onset of the stroke
Change in Motricity index from initial evaluation to the final evaluation | 8 weeks, 12 weeks, 16 weeks from the first onset of the stroke
Change in Functional Oral Intake Scale (FOIS) from initial evaluation to the final evaluation | 8 weeks, 12 weeks, 16 weeks from the first onset of the stroke
Change in MMSE from initial evaluation to the final evaluation | 8 weeks, 12 weeks, 16 weeks from the first onset of the stroke

CONTACTS AND LOCATIONS:
Overall Officials: Geun-Young Park, Study Director — Bucheon St. Mary's Hospital; Yongmin Choi, Principal Investigator — Bucheon St. Mary's Hospital; Sun Im, Study Director — Bucheon St. Mary's Hospital
Locations (1):
- Bucheon St. Mary's Hospital, Bucheon-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided